CLINICAL TRIAL: NCT01781403
Title: Preoperative Chemoradiation With Capecitabine Plus Temozolomide in Patients With Locally Advanced Resectable Rectal Cancer: Phase I Study
Brief Title: Preoperative CRT With Temozolomide Plus Capecitabine in Rectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Tae Won Kim, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML28381
Record Dates: First submitted 2013-01-21; First posted 2013-02-01 (Estimated); Results first posted 2016-06-23 (Estimated); Last update posted 2021-02-04 (Actual); Status verified 2021-01

CONDITIONS: Rectal Cancer
Keywords: Temozolomide; capecitabine; rectal cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Temozolomide; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Capecitabine, Temozolomide, Radiotherapy (Experimental): The total dose of radiotherapy will be 50.4 Gy, with a daily dose of 1.8 Gy administered on 5 days of each week, comprising a total of 45 Gy to the whole pelvis, followed by a 5.4 Gy boost to the primary tumor.
  The doses and schedules for capecitabine will be fixed, with only temozolomide being prescribed using a dose-escalation schedule. Capecitabine and temozolomide will be administered during radiotherapy with drug holidays (weekend break).
  Interventions: Drug: Temozolomide

INTERVENTIONS:
Drug: Temozolomide — Preoperative chemoradiotherapy with fixed dose of capecitabine and temozolomide, the dose of temozolomide will be escalated for finding MTD and RD.
  Other Names: Capecitabine, preoperative radiotherapy

SUMMARY:
The investigators planned a phase I study of preoperative CRT with capecitabine plus temozolomide inpatients with locally advanced resectable rectal cancer: 1) the role of temozolomide as a radiosensitizer has been well established, 2) hypermethylation (or low expression) of MGMT promoter is associated with colorectal carcinogenesis, can be found in 20~40% of colorectal cancer patients, and this proportion could be adequate for validation as its role of predictive biomarker, and 3) temozolomide can be additive or synergistic because radiotherapy is now essential in the treatment of rectal cancer.

DETAILED DESCRIPTION:
Preoperative chemoradiation (CRT) with fluoropyrimidine (5-fluorouracil or capecitabine) is now regarded as a standard treatment option in patients with locally advanced resectable rectal cancer, and pathologic response rates and tumor regression grades after preoperative CRT have been proved to be important prognostic factors for survival outcomes. Several studies of preoperative CRT with fluoropyrimidines plus other agents, such as oxaliplatin, irinotecan, cetuximab, and bevacizumab, have been performed to improve pathologic response rates; however, they have failed to show improved results compared to those with fluoropyrimidine alone. Thus, fluoropyrimidine alone is a standard chemotherapeutic strategy in patients with locally advanced resectable rectal cancer who will be treated with preoperative CRT at present; further studies are needed to find effective combination for improving pathologic responses other than fluoropyrimidines alone in these patient population.

Temozolomide is an oral alkylating agent, and has been proved to be effective in patients with glioblastoma or high grade anaplastic glioma when administered with concurrent radiotherapy either as adjuvant or recurrent settings, and also seemed to be effective in patients with malignant melanoma either as monotherapy or combination chemotherapy. Temozolomide has been known to deplete O6-methylguanine DNA methyltransferase (MGMT), which is one of the DNA repair enzymes, and recent studies have shown that lower expression (by immunohistochemistry) or hypermethylation (by methylation-specific PCR) of MGMT could be a predictive marker of better responses to treatment with temozolomide in patient with glioblastoma, high grade anaplastic glioma or malignant melanoma.

Silencing of MGMT by promoter hypermethylation has been known to involve colorectal carcinogenesis pathway by the association with KRAS mutation and low-CIMP (CpG island methylation phenotype), and hypermethylation of MGMT promoter could be detected in 29% to 46% of tumor tissues from sporadic colorectal cancer patients. Nagasaka et al. showed notable results that MGMT promoter methylation status was associated with microsatellite instability and hypermethylation of MGMT promoter could be a predictive factor of low recurrence in colorectal cancer patients with adjuvant oral fluoropyrimidine chemotherapy after curative surgery. In addition, Shacham-Shmueli et al. showed that temozolomide could be an additional treatment option in a small group of patients with chemotherapy-refractory metastatic colorectal cancer which had lower MGMT expressions.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the rectum
* Tumor located within 12cm of anal verge
* Clinical stage of T3-4 or N+ by rectal MRI with or without endorectal ultrasound
* Available tumor samples before study treatment (fresh or paraffin-embedded) for immunohistochemistry (IHC) and methylation-specific PCR (MSP) to investigate MGMT expression and hypermethylation
* Male or female aged over 20 years
* Be ambulatory and have an Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* No prior systemic treatment (chemotherapy, immunotherapy) or radiation therapy
* Adequate major organ functions as following:
* Be willing and able to comply with the protocol for the duration of the study.
* Give written informed consent prior to study-specific screening procedures, with the understanding that the patient has the right to withdraw from the study at any time, without prejudice.

Exclusion Criteria:

* Histology other than adenocarcinoma or tumor arising from inflammatory bowel disease
* Inadequate tumor sample for MGMT IHC or MSP
* Any evidence of systemic metastasis
* Unresected synchronous colon cancer
* Intestinal obstructions or impending intestinal obstruction, but bypass surgery (colostomy or ileostomy) is permitted before study treatment
* Uncontrolled or severe cardiovascular disease
* Serious concurrent infection or nonmalignant illness that is uncontrolled or whose control may be jeopardized by complications of study therapy.
* Other malignancy within the past 5 years except cured non-melanomatous skin cancer, carcinoma in situ of the cervix, or thyroid papillary carcinoma.
* Organ allografts requiring immunosuppressive therapy.
* Psychiatric disorder or uncontrolled seizure that would preclude compliance.
* Pregnant, nursing women or patients with reproductive potential without contraception.
* Patients receiving a concomitant treatment with drugs interacting with 5-FU such as flucytosine, phenytoin, or warfarin et al.
* Known dihydropyrimidine dehydrogenase (DPD) deficiency.
* Known hypersensitivity to any of the components of the study medications.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-05-10 (Actual); Primary Completion 2014-09-03 (Actual); Study Completion 2016-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tae Won Kim, Professor, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Songpa-gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jeong JH, Hong YS, Park Y, Kim J, Kim JE, Kim KP, Kim SY, Park JH, Kim JH, Park IJ, Lim SB, Yu CS, Kim JC, Kim TW. Phase 1 Study of Preoperative Chemoradiation Therapy With Temozolomide and Capecitabine in Patients With Locally Advanced Rectal Cancer. Int J Radiat Oncol Biol Phys. 2016 Oct 1;96(2):289-295. doi: 10.1016/j.ijrobp.2016.05.009. Epub 2016 May 17. PMID 27473815

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 14 May 2013 through 8 May 2014
Groups:
- Capecitabine 825mg/m^2, Temozolomide 45mg/m^2, Radiotherapy; Capecitabine 825mg/m^2, Temozolomide 60mg/m^2, Radiotherapy; Capecitabine 825mg/m^2, Temozolomide 75mg/m^2, Radiotherapy: The total dose of radiotherapy will be 50.4 Gy, with a daily dose of 1.8 Gy administered on 5 days of each week, comprising a total of 45 Gy to the whole pelvis, followed by a 5.4 Gy boost to the primary tumor.
  The doses and schedules for capecitabine will be fixed, with only temozolomide being prescribed using a dose-escalation schedule. Capecitabine and temozolomide will be administered during radiotherapy with drug holidays (weekend break).
  Temozolomide: Preoperative chemoradiotherapy with fixed dose of capecitabine and temozolomide, the dose of temozolomide will be escalated for finding MTD and RD.
Period: Overall Study
Arm/Group | Capecitabine 825mg/m^2, Temozolomide 45mg/m^2, Radiotherapy | Capecitabine 825mg/m^2, Temozolomide 60mg/m^2, Radiotherapy | Capecitabine 825mg/m^2, Temozolomide 75mg/m^2, Radiotherapy
Started | 2 | 2 | 18
Completed | 2 | 2 | 18
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Capecitabine, Temozolomide, Radiotherapy: The total dose of radiotherapy will be 50.4 Gy, with a daily dose of 1.8 Gy administered on 5 days of each week, comprising a total of 45 Gy to the whole pelvis, followed by a 5.4 Gy boost to the primary tumor.
  The doses and schedules for capecitabine will be fixed, with only temozolomide being prescribed using a dose-escalation schedule. Capecitabine and temozolomide will be administered during radiotherapy with drug holidays (weekend break).
  Temozolomide: Preoperative chemoradiotherapy with fixed dose of capecitabine and temozolomide, the dose of temozolomide will be escalated for finding MTD and RD.
Arm/Group | Capecitabine, Temozolomide, Radiotherapy
Number analyzed (Participants) | 22
Age, Continuous [Median (Full Range); unit: years] | 54 [41 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 15
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 22

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: The MTD is defined as the maximum dose level in the doses of temozolomide tested with capecitabine and radiation in which the incidence proportion of DLT exceeds 30%.
Time Frame: 5-6 weeks during study treatment
Measure: Number; unit: mg/m^2
Groups:
- Dose Level 1: Capecitabine was given 825 mg/m^2 twice/day during radiotherapy with drug holidays (weekend breaks).
  Temozolomide was given 45 mg/m^2 once/day during radiotherapy with drug holidays (weekend breaks).
- Dose Level 2: Capecitabine was given 825 mg/m^2 twice/day during radiotherapy with drug holidays (weekend breaks).
  Temozolomide was given 60 mg/m^2 once/day during radiotherapy with drug holidays (weekend breaks).
- Dose Level 3/Recommended Dose: Capecitabine was given 825 mg/m^2 twice/day during radiotherapy with drug holidays (weekend breaks).
  Temozolomide was given 75 mg/m^2 once/day during radiotherapy with drug holidays (weekend breaks).
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3/Recommended Dose
Number analyzed (Participants) | 2 | 2 | 18
mg/m^2 | 0 | 0 | 0

2. Primary Outcome: Recommended Dose (RD)
Description: RD will be defined as one level below the MTD.
Time Frame: 5-6 weeks after CRT
Measure: Number; unit: mg/m^2
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3/Recommended Dose
Number analyzed (Participants) | 2 | 2 | 18
mg/m^2 | 0 | 0 | 75

3. Secondary Outcome: Pathological Complete Response
Description: Pathologic responses and stages were classified according to Dworak's classification and the 7th edition of the American Joint Committee on Cancer staging system, respectively.
  The pathologic complete response (pCR) was defined as the total regression of the primary tumor regardless of regional lymph nodal status (ypT0), with residual fibrotic mass or acellular mucin pools only, thus without detectable tumor cells.
Time Frame: at the time of surgery (6-8 weeks after study treatment)
Measure: Number; unit: participants
Groups:
- Unmethylated MGMT: MGMT methylation specific PCR: unmethlyated
- Hypermethylated MGMT: MGMT methylation specific PCR: hypermethylated
Arm/Group | Unmethylated MGMT | Hypermethylated MGMT
Number analyzed (Participants) | 6 | 16
participants | 1 | 6

4. Other Pre Specified Outcome: Toxicity(Adeverse Event)
Description: Toxicity will be monitored and recorded every week during study treatment (5 or 6 weeks) as following according to the NCI-CTCAE version 4.0
  1. An interval history and physical examination with particular attention to drug-induced side effects along with documentation of the patient's weight and performance status will be performed on each visit.
  2. CBC with differential count, blood chemistry including calcium, phosphorus, glucose, BUN, creatinine, total protein, albumin, AST, ALT, alkaline phosphatase, total bilirubin, and electrolyte will be performed before next planned treatment.
  3. All relevant information regarding drug dosage, laboratory examinations, and treatment-related toxicities must be recorded before each treatment is given.
  4. Summaries of the frequency and severity of adverse effects are based on the worst episodes recorded.
Time Frame: 5-6 weeks during study treatment
Measure: Number; unit: events
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3/Recommended Dose
Number analyzed (Participants) | 2 | 2 | 18
events
  Any grade 1 adverse event | 6 | 8 | 60
  Any grade 2 adverse event | 2 | 2 | 17
  Any grade 3 adverse event | 1 | 0 | 3
  Any grade 4 adverse event | 0 | 0 | 0

5. Other Pre Specified Outcome: Efficacy: Pathologic Major Responses
Description: Efficacy: Pathologic major responses = total regression + near total regression.
  We will carefully inspect the circumferential resection margin, defining a positive margin as any residual tumor within ≤ 1 mm of the circumferential margin.
  Pathologic responses and stages will be classified according to Dworak's classification1 and the AJCC (American Joint Committee on Cancer) staging system, respectively. In each case, the entire tumor including mesorectal fat will be serially sliced into 4-mm-thick sections and embedded in paraffin.
  A pathologic complete response is defined as grade 4 tumor regression; with residual fibrotic mass or acellular mucin pools only, thus without detectable tumor cells
  A near total response is defined as grade 3 tumor regression; with very few tumor cells in fibrotic tissue with or without mucous substance.
Time Frame: after surgery (6-8 weeks after study treatment)
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Disease-free Survival
Time Frame: 3-year or 5-year after surgery
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3/Recommended Dose
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/18
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2 | 18/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=2) | Dose Level 2 (N=2) | Dose Level 3/Recommended Dose (N=18)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 10 (10)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 13 (13)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 7 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 4 (4)
Anorexia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 6 (6)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 14 (14)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 5 (5)
Fatigue (General disorders) | 1 (1) | 2 (2) | 3 (3)
Hand-foot syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0)
ALT abnormalities (Hepatobiliary disorders) | 0 (0) | 0 (0) | 7 (7)
AST abnormalities (Hepatobiliary disorders) | 0 (0) | 0 (0) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other